CLINICAL TRIAL: NCT01762449
Title: Morbidity and Mortality Follow Up of Participants of the Scleroderma Lung Study 1
Brief Title: Morbidity and Mortality Follow Up for the Scleroderma Lung Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00026357
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Scleroderma
Keywords: Scleroderma; interstitial lung disease
MeSH Terms: conditions — Scleroderma, Diffuse; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients who received cyclophosphamide: Patients who received cyclophosphamide on the Scleroderma Lung Study
  Interventions: Other: Followup survey
- Patients who received placebo: Patients who received placebo on the Scleroderma Lung Study
  Interventions: Other: Followup survey

INTERVENTIONS:
Other: Followup survey

SUMMARY:
The primary intent of this study is to add to the body of knowledge on scleroderma patients with interstitial lung disease. While lung disease is recognized as the leading cause of death amongst patients with scleroderma, there is not a large body of literature describing the long-term morbidity and mortality rate of these scleroderma patients. For this reason, the investigators are following participants of the Scleroderma Lung Study (NCT00004563) after their participation in that study was concluded. In addition, the investigators will assess if the subjects who received one year of oral cyclophosphamide in the Scleroderma Lung Study experienced progression of their scleroderma-related lung disease following the end of the study.

DETAILED DESCRIPTION:
Retrospective and prospective data will be collected about patients who participated in the Scleroderma Lung Study (SLS). An attempt will be made to include all of the participants of the Scleroderma Lung Study, who were reported as alive at the end of that study.

A total of 158 subjects (79 per treatment arm) were randomized on the original Scleroderma Lung Study. Of those, 109 subjects completed the study. A single telephone interview with the participants to assess the occurrence of severe events and a review of the participant's medical records may be conducted. The outcome information will be combined with information collected about all participants in the SLS study. The data being collected includes information on mortality, development of cancers, development of organ failure, and performance status.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the Scleroderma Lung Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who participated in the Scleroderma Lung Study
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Time to death or first organ failure | 9-12 years

CONTACTS AND LOCATIONS:
Overall Officials: Keith Sullivan, MD, Study Chair — Duke University; Daniel Furst, MD, Study Chair — University of California, Los Angeles; Donald Tashkin, MD, Principal Investigator — University of California, Los Angeles